CLINICAL TRIAL: NCT04955522
Title: Multimodal Imaging Analysis of Spinal Tumors
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019501
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2019-12

CONDITIONS: Bone Tumor
MeSH Terms: conditions — Bone Neoplasms | interventions — Radiomics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- metastases: patients with spinal metastases
  Interventions: Diagnostic Test: radiomics
- multiple myeloma: patients with spinal multiple myeloma

INTERVENTIONS:
Diagnostic Test: radiomics — Differential diagnosis of spinal myeloma and metastases by radiomics
  Groups: metastases

SUMMARY:
In this study, we retrospectively analyzed the imaging data of spinal tumors to find out more imaging features of spinal tumors, in order to provide more accurate reference for the diagnosis of spinal tumors.

DETAILED DESCRIPTION:
Bone tumors account for 1-2% of total body tumors, and spinal tumors only account for 6.5% of total body tumors. Because of the low incidence rate, the number of patients and the attention in this field are far lower than other tumors, so far, all the researches on spinal tumors are relatively lacking. Because the diagnosis of bone tumor needs the combination of clinical, imaging and pathological to make a more accurate diagnosis, so the imaging diagnosis of spinal tumor is very important. In this study, through retrospective analysis of a variety of imaging data of patients with spinal tumor, measurement and recording of spinal tumor image related parameters, and statistical analysis, in order to find out more imaging characteristics of patients with spinal tumor, more accurate diagnosis of lesions, and provide more help for clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Complete and accurate clinical and pathological data are available；Imaging examination was performed in our hospital

Exclusion Criteria:

* Patients with missing image data and unclear image

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Spinal tumor patients in Peking University Third Hospital from January 2006 to October 2019
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
radiomics features | 2020.12.1-2020.12.25
  1409 radiomics features can be extracted from the images. Objective to search for the radiomics index which is helpful to the diagnosis of tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Huishu Yuan, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China